CLINICAL TRIAL: NCT02967796
Title: Descriptive Study About a Strategy of Micronutrient Management in Parturient and Layered Women With Proteochoc®, a Dietary Supplement Rich in Porphyra HSP®
Brief Title: Strategy of Micronutrient Management in Parturient and Layered Women With a Dietary Supplement Rich in Porphyra HSP®
Status: Completed | Type: Observational
Sponsor: PiLeJe (Industry)
Responsible Party: Sponsor
Other Study IDs: PiL-Obs-ProtSC-014
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Postpartum Perineal Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Supplemented group: 6 capsule of Proteochoc during 4 day, from day 0 (day of delivery) to day 4
  Interventions: Dietary Supplement: Proteochoc
- Control group: no supplementation, just the same follow-up as supplemented group

INTERVENTIONS:
Dietary Supplement: Proteochoc
  Groups: Supplemented group

SUMMARY:
The aim of the study is to evaluate in primiparous patients the benefit of supplementation with Proteochoc® to reduce perineal pain in the postpartum especially, in sitting posture. The patient is followed from the delivery to 6 to 8 weeks after.

DETAILED DESCRIPTION:
For this study, 60 patients are going to be included. There will be 2 groups : a supplemented one (proteochoc®) and a non supplemented one (control). The patients of these two groups will have the same follow-up At the time of inclusion, an inclusion card is completed describing the patient's socio-demographic characteristics, major medical, surgical and obstetric history. After an uncomplicated delivery, women stay in maternity for a maximum of 3 days. In accordance with standard medical practice, women will be seen daily from D0 to D + 3 by the nursing staff. The investigating physician and his team will complete the follow-up sheets in the aftermath (day1), day3 and 6-8 weeks after the usual visits.

The data collected are information on medication treatments, prescribed care, assessment of the patient's overall condition and recovery, and monitoring of perineal lesions and complications if applicable.

In the same time (day1, day3, day6, day14 and 6-8 weeks after, the patient will also complete a patient follow-up sheet to collect her impressions.

The data collected are the medications taken, the care taken, the general pain felt, the perineal pain felt if applicable, and the fatigue felt.

ELIGIBILITY:
Inclusion Criteria:

* Female aged over 18
* First pregnancy
* Having given birth, at a term greater than or equal to 37 SA, by low route, of a single child born alive and not hospitalized in the aftermath of immediate layers
* For whom the investigator has freely decided to propose a complementation by Protéochoc® on the day of delivery and its sequences of layers
* Having freely decided to buy Protéochoc® and follow the advice of consumption proposed by its gynecologist-obstetrician
* Having agreed to sign a consent to participate in the investigation after receiving informed information from the investigator

Exclusion Criteria:

* Serious pathology running
* Suffering before the pregnancy of any of the following conditions:
* Chronic pelvic pain syndrome
* Ilio-inguinal, ilio-hypogastric and genito-femoral pudendal neuralgia
* Pains with osteo-ligamentary component: the syndrome of the dorsolumbar hinge and the coccygodynia
* Myofacial Syndrome
* Pain of muscular origin: the syndrome of the pyriform muscle, syndrome of the obturator muscle
* Pains of venous origin: pelvic varices
* Allergy to any of the components of Proteochoc®
* Patient refusing to participate or unable to participate in the survey due to major language problems or major neuropsychiatric disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women running their first pregnancy
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-09-04 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

PRIMARY OUTCOMES:
perineal pain intensity in the sitting position | day 6
  The primary outcome will be the perineal pain intensity in the sitting position measured by a visual analogue scale (rated 0 to 10) at day 6 in women who chose to complement versus women who did not wish to take the supplementation

SECONDARY OUTCOMES:
Doctor's evaluation | Day 1 (day after the delivery)
  Taking other medication Prescription of perineal care General condition of the patient Post-delivery recovery Type of perineal lesion and its evolution if applicable Complications and their evolutions if applicable Evolution of the scar(s) of the tear(s) or episiotomy if applicable Compliance with the Protéochoc® product
Doctor's evaluation | Day 3
  Taking other medication Prescription of perineal care General condition of the patient Post-delivery recovery Type of perineal lesion and its evolution if applicable Complications and their evolutions if applicable Evolution of the scar(s) of the tear(s) or episiotomy if applicable Compliance with the Protéochoc® product
Doctor's evaluation | Day 56
  Taking other medication Prescription of perineal care General condition of the patient Post-delivery recovery Type of perineal lesion and its evolution if applicable Complications and their evolutions if applicable Evolution of the scar(s) of the tear(s) or episiotomy if applicable Compliance with the Protéochoc® product
Patient's evaluation | Day 1 (day after the delivery)
  Taking other medication Perineal care performed The level of pain in general, uterine pain and breast pain The level of perineal pain and its evolution The discomfort caused by perineal pain (rest, walking and urination) The state of fatigue (fatigue score, score 0 to 4) Compliance with the Protéochoc® product
Patient's evaluation | Day 3
  Taking other medication Perineal care performed The level of pain in general, uterine pain and breast pain The level of perineal pain and its evolution The discomfort caused by perineal pain (rest, walking and urination) The state of fatigue (fatigue score, score 0 to 4) Compliance with the Protéochoc® product
Patient's evaluation | Day 6
  Taking other medication Perineal care performed The level of pain in general, uterine pain and breast pain The level of perineal pain and its evolution The discomfort caused by perineal pain (rest, walking and urination) The state of fatigue (fatigue score, score 0 to 4) Compliance with the Protéochoc® product
Patient's evaluation | Day 14
  Taking other medication Perineal care performed The level of pain in general, uterine pain and breast pain The level of perineal pain and its evolution The discomfort caused by perineal pain (rest, walking and urination) The state of fatigue (fatigue score, score 0 to 4) Compliance with the Protéochoc® product
Patient's evaluation | Day 56
  Taking other medication Perineal care performed The level of pain in general, uterine pain and breast pain The level of perineal pain and its evolution The discomfort caused by perineal pain (rest, walking and urination) The state of fatigue (fatigue score, score 0 to 4) Compliance with the Protéochoc® product

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier d'Auch, Auch, France